CLINICAL TRIAL: NCT05665361
Title: A Phase I/II Study of Palbociclib and Sasanlimab for the Treatment of Advanced Clear Cell Renal Cell Carcinoma (ccRCC) or Papillary Renal Cell Carcinoma (pRCC)
Brief Title: Palbociclib and Sasanlimab for the Treatment of Advanced Clear Cell Renal Cell Carcinoma (ccRCC) or Papillary Renal Cell Carcinoma (pRCC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000666; 000666-C
Record Dates: First submitted 2022-12-23; First posted 2022-12-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Advanced Clear Cell Renal Carcinoma (Ccrcc); Papillary Renal Cell Carcinoma (Prcc)
Keywords: Papillary Renal Cell Carcinoma; Kidney Neoplasms; Kidney Cancer; Clear Cell Renal Cell Carcinoma; Translocation Renal Cell Carcinoma; TFE3-rearranged renal cell cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Phase I (Experimental): Sasanlimab and deescalating doses of palbociclib
  Interventions: Drug: Sasanlimab; Drug: Palbocicilib
- 2/Phase II (Experimental): Sasanlimab and palbociclib at the dose determined in Phase I (RP2D)
  Interventions: Drug: Sasanlimab; Drug: Palbocicilib

INTERVENTIONS:
Drug: Sasanlimab — Sasanlimab will be given (SC on day 1 of every cycle, starting on day 1 (+/- 5 days) of cycle 2).
Drug: Palbocicilib — Palbociclib will be given PO for 21 days of every 28-day cycle, starting on day 1 of cycle 1.

SUMMARY:
Background:

Kidney cancer is the 12th leading cause of cancer-related death in the United States. Some kidney tumors do not respond well to current treatments. Better treatments are needed.

Objective:

To test a pair of drugs (sasanlimab and palbociclib) in people with kidney cancers.

Eligibility:

People aged 18 years and older with kidney cancer; specifically, clear cell renal cell carcinoma (ccRCC) or papillary renal cell carcinoma (pRCC).

Design:

Participants will be screened. They will have a physical exam with blood tests. They will have an imaging scan and a test of their heart function. They may have a biopsy; that is, a sample of tissue will be cut from the tumor.

Participants will be treated in 28-day cycles for up to 2 years.

Palbociclib is a pill taken by mouth. Participants will take this drug once a day for 21 days during each 28-day treatment cycle. They will write down the dates and times they take these pills in a diary.

Sasanlimab is an injection under the skin. Participants will receive this injection on the first day of each treatment cycle.

Imaging scans and blood tests will be repeated throughout the treatment. Tumor biopsies may be repeated up to 3 times; these biopsies are optional.

Participants will have follow-up visits every month for 3 months after treatment ends. They will continue to have imaging scans every 3 months; these scans may be done close to home. The results can be sent to researchers.

Participants will remain in the study up to 6 years.

DETAILED DESCRIPTION:
Background:

* Kidney cancer is the 8th most common malignancy and 12th leading cause of cancer-related death in the United States. It is estimated that there will be 79,000 new cases of kidney cancer diagnosed in 2022, resulting in 13,920 deaths. Despite a steady increase in the incidence of renal cell cancer (RCC) over the past 3 decades, there has been an improvement in observed 5-year survival rates.
* Most patients with advanced clear cell RCC are treated with immune checkpoint inhibitors targeting the programmed cell death protein 1 (PD-1) and/or the CTLA4 axis and agents targeting the vascular endothelial growth factor (VEGF) pathway. There is a paucity of options for patients who have progressed on these therapies. There is currently no widely accepted standard for patients with papillary RCC, although some patients may benefit from agents such as cabozantinib or the combination of bevacizumab and erlotinib.
* Preclinical data suggest that inhibitors of CDK 4/6 might be active in kidney cancer and that these agents might act synergistically with PD-1 checkpoint inhibitors in a variety of preclinical models.
* Palbociclib is a highly selective, reversible oral inhibitor of cyclin-dependent kinases (CDK) 4 and 6. Inhibition of CDK 4/6 blocks DNA synthesis by prohibiting the progression of the cell cycle from G1 to the S phase. Data from nonclinical studies indicate that palbociclib may have cytostatic effects on tumor cells.
* Sasanlimab is an investigational humanized immunoglobulin G4 monoclonal antibody that binds PD-1 and blocks its interaction with its ligands, programmed death-ligand 1 and 2 (PD-L1) & (PD-L2). It presents the distinct characteristic that it can be administered subcutaneously on a monthly basis whereas approved and other available anti-PD-1/PDL1 therapies currently are administered intravenously. In animal models, it demonstrated high-affinity interaction with PD 1 and was associated with a significant delay in the growth of murine MC-38 colorectal tumors implanted in hu-PD-1 knock-in mice.

Objectives:

* Phase I: To determine recommended phase II dose (RP2D) of palbociclib in combination with sasanlimab
* Phase II: To determine the overall response rate (ORR) defined as partial response (PR) + complete response (CR) of the RP2D of the combination of palbociclib and sasanlimab in participants with advanced ccRCC (Cohorts 1a and 2a) and advanced pRCC (Cohorts 1b and 2b) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

Eligibility:

* Age 18 years or older
* Participants with histologically or cytologically confirmed advanced ccRCC or pRCC
* Participants must have measurable disease per RECIST 1.1
* ECOG performance status <= 1
* Adequate organ function as defined by the liver, kidney, and hematologic laboratory testing
* Participants with ccRCC must have received checkpoint inhibitor therapy and must have received or been ineligible to receive a VEGF pathway antagonist (as a single agent or as part of a combination)
* Participants with pRCC can be treatment-na(SqrRoot) ve or have previously received systemic treatment for pRCC.
* No more than four prior lines of therapy in the metastatic setting.

Design:

* The proposed study is an open label, phase I/II study of palbociclib in combination with sasanlimab
* Participants will be enrolled simultaneously into Cohort 1a (ccRCC) and Cohort 1b (pRCC) and start treatment in cycles consisting of 28 (+/- 5) days
* Initially, 6-18 participants from Cohort 1a and/or Cohort 1b will be enrolled into Phase I to estimate RP2D. If RP2D is estimated, we will continue enrollment as planned into Phase II, if not, we will submit amendment with updated dosing
* Following the Phase I, the first 9 participants from each pair of Cohorts (1a+2a) and (1b+2b) enrolled at the RP2D of palbociclib and sasanlimab in Phase I and Phase II will be evaluated separately for response. If among these 9 participants from pair of Cohorts (1a+2a) and (1b+2b), no more than 1 objective response defined as CR+PR is seen, then no further participants will be enrolled in Cohort 2a or 2b

ELIGIBILITY:
* INCLUSION CRITERIA:
* Cytologically or histologically confirmed clear cell renal cell carcinoma (presence of a clear cell component) (ccRCC) (Cohort 1) or papillary renal cell carcinoma (pRCC) (presence of a papillary component) (Cohort 2)
* Participants must have advanced RCC with at least one measurable lesion as outlined in RECIST 1.1.
* Participants with ccRCC (Cohort 1) must have received checkpoint inhibitor therapy and must have received or been ineligible to receive a VEGF pathway antagonist (as a single agent or as part of a combination)
* Participants with pRCC (Cohort 2) can be treatment-na(SqrRoot) ve or have previously received systemic treatment for pRCC
* Age >= 18 years
* ECOG performance status <= 1
* Adequate hematologic function at screening, as follows:

  * Absolute neutrophil count (ANC) >= 1,000/microliter
  * Hemoglobin (Hb) >= 9 g/dL with no blood transfusion within 2 weeks prior to treatment initiation
  * Platelets >= 100,000/microliter
* Adequate renal and hepatic function at screening, as follows:

  * Serum creatinine <= 1.5 x upper limit of normal (ULN) OR, if >1.5x ULN, creatinine clearance (CrCl) >= 30 mL/min/1.73 m^2 (calculated CrCl (CKD-EPI or calculated eGFR provided by laboratory))
  * Total bilirubin <= 1.5 x ULN OR in participants with known or suspected Gilbert's syndrome, total bilirubin <= 3.0 x ULN
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2.5 x ULN, (unless liver metastases are present, then values must be <= 5 x ULN)
* Participants serologically positive for hepatitis C virus (HCV) are eligible if HCV viral load is undetectable
* Participants serologically positive for human immunodeficiency virus (HIV) are eligible if they are on stable antiretroviral therapy for at least 4 weeks before treatment initiation, have no reported opportunistic infections or Castleman s disease within 12 months prior to treatment initiation, have a viral load that is undetectable by quantitative polymerase chain reaction (PCR) and CD4 count >= 200 cells per cubic millimeter
* Participants with brain metastasis are eligible if at least 4 weeks status post radiotherapy or surgery before treatment initiation with no evidence of progression or associated symptoms
* Women of child-bearing potential (WOCBP) must agree to use one (1) highly effective method of contraception (e.g.,hormonal, intrauterine device (IUD), surgical sterilization) prior to study entry, for the duration of study therapy, and for up to 6 months following the last dose of any study agent(s). Women must refrain from donating eggs during this same period. NOTE: WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.
* Men with female partners of reproductive potential and pregnant partners are required to use a condom (even after vasectomy), during treatment and for at least 6 months after the final dose and must refrain from donating sperm during this same period.
* Breastfeeding participants must be willing to discontinue breastfeeding from study enrollment through 6 months after study treatment discontinuation
* Participants must be able to understand and be willing to sign a written informed consent document

EXCLUSION CRITERIA:

* Prior treatment for RCC with chemotherapy, hormonal therapy, immunotherapy, treatment with an experimental agent, and/or radiation therapy within 4 weeks or 5 halflives, whichever is shorter, prior to treatment initiation
* More than four prior lines of systemic therapy in the metastatic setting
* Participants who have wound dehiscence from prior surgeries
* Active inflammatory bowel disease, chronic diarrhea, gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of palbociclib
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study agents
* Prior history of grade >=3 immune-related adverse event(s) with checkpoint inhibitor therapy. Note: participants who had endocrine toxicity of grades 3 or 4 are eligible
* An active autoimmune disease. Note: participants with type 1 diabetes, eczema, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease, adrenal insufficiency on systemic oral corticosteroid therapy (<= the equivalent of prednisone 10 mg/day) or other mild autoimmune disorders not requiring immunosuppressive treatment are eligible.
* Participants receiving systemic corticosteroids at doses equivalent > 10 mg/daily of prednisone, cyclophosphamide, azathioprine, methotrexate, mycophenolate mofetil, sirolimus, thalidomide, or anti-tumor necrosis factor [anti-TNF] agents. Note: participants on steroids through a route known to result in minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are eligible
* Prior allogeneic/autologous bone marrow or solid organ transplant
* Participants with current or past hepatitis B (HBV) infection
* Participants with a history of interstitial lung disease, non-infectious pneumonitis, or untreated active/latent pulmonary tuberculosis (TB)
* Participants taking medications that are strong inhibitors or inducers of CYP3A (https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-druginteractions-table-substrates-inhibitors-and-inducers#table3-2) within 21 days or 5 half-lives of the agent (whichever is shorter) prior to initiation of study therapy
* Participants taking any herbal supplements within 14 days prior to initiation of study therapy
* History of a non RCC malignancy within 2 years of treatment initiation except for the following: adequately treated localized skin cancer, ductal carcinoma in situ, cervical carcinoma in situ, superficial bladder cancer, or other malignancy which does not require treatment at the current time per Standard of Care
* Pregnant women (confirmed by beta-HCG serum pregnancy test performed at screening)
* Uncontrolled intercurrent illness that would limit compliance with study requirements, evaluated by history, physical exam, and chemistry panel.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: To determine RP2D of palbociclib in combination with sasanlimab | 28 days
  Number of DLTs within DLT period
Phase II: Objective response rate (ORR) | 6 years
  Responses (PR+CR) in participants based on imaging [CT scan of chest, abdomen, and pelvis (or MRI of abdomen and pelvis with CT chest without contrast when appropriate)] performed every 8 (+/-1) weeks for 32 weeks and every 12 (+/-1) weeks after that until the first of either disease progression or 6 years after enrollment

SECONDARY OUTCOMES:
Disease Control Rate (DCR) defined as PR + CR+ SD in participants re-treated with the study drug combination by RECIST 1.1 | 6 years
  DCR as assessed by imaging [CT scan of chest, abdomen, and pelvis (or MRI of abdomen and pelvis with CT chest without contrast when appropriate)] performed every 8 (+/-1) weeks for 32 weeks and every 12 (+/-1) weeks after that until the first of either disease progression or 6 years after enrollment
progression-free survival (PFS) | 6 years
  Progression free survival determined by imaging [CT scan of chest, abdomen, and pelvis (or MRI of abdomen and pelvis with CT chest without contrast when appropriate)] performed every 8 (+/-1) weeks for 32 weeks and every 12 (+/-1) weeks after that until the first of either disease progression or 6 years after enrollment
safety of the combination of palbociclib and sasanlimab | 6 years
  Any toxicities identified between Day 1 of Cycle 1 through 90 days after the study agent (s) was/were last administered will be collected and reported by type and grade. Beyond 90 days after the last intervention, only adverse events which are serious and related to the study intervention will be recorded and reported. Note: during re-treatment AEs will be documented from the re-start of the study intervention through 90 days after the study agent (s) was/were last administered. Beyond 90 days after the last intervention, only adverse events which are serious and related to the study intervention need to be recorded
overall survival (OS) | 6 years
  Participants assessed at Day 1 of every cycle, safety follow up visits at days 30, 60, 90, every 12 weeks until progression and/or every 6 months after progression for 6 years after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Ramaprasad Srinivasan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All large scale genomic sequencing data will be shared with subscribers to dbGaP. All collected IPD will be shared with other investigators after publication in accordance with the executed CRADA.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested by other researchers at the time of publication or shortly thereafter. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active
Access Criteria: Data from this study may be requested by contacting the PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000666-C.html